CLINICAL TRIAL: NCT05233423
Title: The Effect of Pressurized Cold Application on Pain Level in Patients Wıth Total Knee Prosthesis Surgery
Brief Title: Pressurized Cold Application for Patients Total Knee Prosthesis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Özge Buldan, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OBuldan
Record Dates: First submitted 2021-12-28; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-12

CONDITIONS: Knee Prosthesis; Cryotherapy; Pain; Patient Satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The patients in the intervention group were applied 9 cold applications with 30 mmHg pressure for 20 minutes and 40 minutes of rest.
  Interventions: Device: compressed cold therapy bandage
- Control Group (No Intervention): The patients in the control group were applied 9 times of cold gel in the form of 20 minutes of application and 40 minutes of rest after surgery.

INTERVENTIONS:
Device: compressed cold therapy bandage — Compressed cold therapy bandage was applied by wrapping the operated knee of the patients. The patients in the intervention group received 9 cold applications with 30 mmHg pressure for 20 minutes and 40 minutes of rest.
  Arms: Intervention Group

SUMMARY:
This study was conducted to examine the effects of pressurized cold applicatıon for patients total knee prosthesis surgery.

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled experimental study in order to determine the effect of pressurized cold application applied after total knee replacement surgery on the level of pain and satisfaction.This study was conducted in 52 patients who applied to Pamukkale University Hospitals Orthopedics and Traumatology Clinic between July 2019 and February 2020, who met the inclusion criteria and accepted to participate in the study. The patients were divided into 26 in the control group (cold gel) and 26 in the study group (compressed cold therapy bandage) using a simple randomization method. The patients in the control group received 9 cold applications, in the form of 20 minutes of application and 40 minutes of rest after surgery. The patients in the study group were applied 9 cold applications with 30 mmHg pressure for 20 minutes and 40 minutes of rest.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* TDP surgery is planned to be performed by the same physician according to the rapid recovery protocol
* volunteer to participate in research
* had no problems in communicating cognitively, emotionally and verbally were included.

Exclusion Criteria:

* have a cold allergy
* have peripheral vascular disease
* diagnosed with Raynaud's disease
* have cognitive, affective and verbal communication problems

Ages: 46 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The change in pain level of total knee prothesis patients at 9 cold applicatiıon with Visual Analog Scale. | According to the fast track protocol, a total of 9 cold applications were applied to the patients who stayed in the service for an average of 1 day after the operation, except during sleep and physical therapy times.
  This scale was used horizontally before and after 9 cold applications to measure the pain level of the patients.

SECONDARY OUTCOMES:
The level of satisfaction of patients with the type of cold application applied | ,The patient was asked once before discharge (about 1 day after surgery), the level of satisfaction with the type of cold application.
  Satisfaction of the patients with the type of cold application applied was evaluated with a 4-point Likert question before discharge. (Very Satisfied, Satisfied, Neutral, Dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No